CLINICAL TRIAL: NCT03907306
Title: Cold Argon Plasma Application in the Wound Treatment After Open Hemorrhoidectomy
Brief Title: Cold Argon Plasma (CAP) Application in the Wound Treatment After Open Hemorrhoidectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120
Record Dates: First submitted 2019-03-22; First posted 2019-04-08 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Cold Argon Plasma
Keywords: Cold argon plasma; hemorrhoidectomy; wound healing; hemorrhoids
MeSH Terms: conditions — Hemorrhoids | interventions — Wound Healing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients after open hemorrhoidectomy (study group) (Experimental): Patients to whom during a post-operation period cold argon plasma and a standard treatment will be treated. Cold argon plasma will be applied during 4 minutes at one session on the 2nd, 3rd, 4th, 5th, 6th, 7th, 8th, 14th, 21nd, 30th day after operation. The usage of antibacterial and wound healing ointments daily.
  Interventions: Procedure: Wound healing
- Patients after open hemorrhoidectomy (control group) (Active Comparator): Patients who during a post-operation period will be treated with a standard treatment.The usage of antibacterial and wound healing ointments daily.
  Interventions: Procedure: Wound healing

INTERVENTIONS:
Procedure: Wound healing — The measurement of a wound area is committed on the 2nd, 8th, 14th, 21nd and 30th day after operation. By means of the mathematical formulas the wound healing speed will be defined. The wound process will be researched with the help of cytological method. The wound prints will be taken on the 2nd, 8th, 14th, 21nd and 30th day after operation. Microbiological research of a wound will be held on the 2nd, 8th, 14th, 21nd and 30th day after operation (in study groups before and after the usage of CAP, in control groups once). The pain assessment will be measured by a visual analogue scale on the 2nd, 3rd,4th, 5th, 6th, 7th, 8th, 14th, 21nd and 30th day after operation. The life quality will be researched by means of Health Status Survey on the 8th and 30th day before operation.

SUMMARY:
This is single-center, prospective, randomized study

DETAILED DESCRIPTION:
This study will include patients with 3-4 stage hemorrhoids. They will undergo an operation of open hemorrhoidectomy. Patients will be divided into a study group and a control group. Study group patients during a post-operation period except a standard treatment (antiseptic solutions and antibacterial and wound healing ointments) of a post-operation wound will be treated with cold argon plasma. Control group patients will be treated with a standard treatment. Wound healing speed will be researched.

ELIGIBILITY:
Inclusion Criteria:

* 3-4 stage hemorrhoids
* 3 hemorrhoids

Exclusion Criteria:

* patients underwent anal canals intervention
* acute hemorrhoids
* inflammatory bowel disease
* co-morbidity diseases of anal canal and perianal area
* concurrent conditions in the stage of decompensation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Wound healing | 30 days
  Total wound healing will be assessed with the help of cytological and macroscopic methods.In the cytological method the presence of fibroblasts, mature epithelial cells, scar tissue formation and the absence of inflammation will be the criterion of wound healing, as well as the presence of macroscopic features of wound epithelialization.

SECONDARY OUTCOMES:
Pain Intensity Measure | 2, 3, 4, 5, 6, 7, 8, 14, 21, 30 days
  Visual analogue scale (0-10 points)
Life quality | before operation, 8 days, 30 days
  Short Form - 36 Health Status Survey
Microbiological contamination of wound area | 2, 8, 14, 21, 30 days
  Microbiological contamination from the post operation wound area. The assessment of CAP effect on bacteria in planktonic and biofilm forms. Microbiological research of a wound will be held on the 2nd, 8th, 14th, 21nd and 30th day after operation (in study groups before and after the usage of CAP, in control groups once).

CONTACTS AND LOCATIONS:
Locations (1):
- State Scientific Centre of Coloproctology, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No